CLINICAL TRIAL: NCT01318343
Title: Analysis of CoolSculpting by Zeltiq for Non-Invasive Cooling of Subcutaneous Fat of the Abdomen Using the eZ App Large Applicator
Brief Title: Analysis of CoolSculpting by Zeltiq for Non-Invasive Cooling of Abdominal Fat Using the eZ App Large Applicator
Status: Completed | Type: Observational
Sponsor: Laser and Skin Surgery Center of New York (Other)
Collaborators: Zeltiq Aesthetics (Industry)
Responsible Party: Roy G. Geronemus, M.D., Laser & Skin Surgery Center of New York
Other Study IDs: LSSC Zeltiq eZ App 8
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Abdominal Fat; Adipose Tissue, Abdominal
Keywords: Cryolipolysis; Abdominal Fat; Adipose Tissue; Fat Reduction; Non Invasive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Treatment Group 1: Eight (8) subjects will receive one (1) treatment with the eZ8 Large Applicator.
- Treatment Group 2: Eight (8) subjects will receive two (2) treatments two (2) months apart with the eZ8 Large Applicator.
- Treatment Group 3: Four (4) subjects will receive one (1) treatment, six (6) months after the previous treatment with the eZ App 8 large applicator to the abdomen. This is the same applicator that is being evaluated in this study. These subjects have been treated on-site at the Laser & Skin Surgery Center of New York by the study doctor.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of single treatment vs. multiple treatments of CoolSculpting™ by Zeltiq™ Aesthetics for non-invasive cooling of subcutaneous fat using the eZ App 8 large applicator on the abdomen for fat layer reduction.

DETAILED DESCRIPTION:
The Zeltiq Cooling Device to be used in this study (i.e, CLN1) is designed to non-invasively cool skin and subcutaneous fat. The device provides cooling at a controlled preset level (i.e., temperature) as defined by a pre-programmed treatment profile and provides continuous feedback on the temperature of the cooling plate interface with the skin. The device also is able to provide warming at a controlled and variable, preset temperature.

The cooling device includes an applicator, which is the component used to apply cooling and warming to the treatment site, and the control unit which houses the system controller, power source, and other hardware. Each applicator is comprised of at least two thermoelectric coolers with an aluminum plate which is the primary skin interface for cooling and warming. The thermoelectric cooler is controlled and powered by a thermoelectric cooler controller is part of the control system. The device allows a well-controlled temperature to be applied to and maintained at the surface of the treatment area.

The Zeltiq Aesthetics Cooling Device to be used in this study has one applicator configuration. The vacuum applicator, which includes a small amount of vacuum pressure to create the massage effect. A disposable sleeve is provided for use with each of these applicators to provide an interface between the applicator and the skin. Sensors are included in the disposable sleeve to measure the temperature at the interface and to provide feedback to ensure appropriate control of the applicator temperature.

For the protection of the subject, safety features are incorporated into the device to avoid any unexpected excursions in the temperature. The device will automatically terminate the procedure if the measured temperature exceeds the minimum and maximum programmed temperature by more than one degree, i.e., 1ºC colder than the minimum programmed cooling temperature or 1ºC warmer than the maximum programmed temperature. Furthermore, the device has been tested extensively prior to being made available for use in this clinical study. Electrical safety tests to established standards (IEC-60601, UL-2601) have been performed and extensive testing has been performed to demonstrate device temperature reproducibility. Biocompatibility testing has been performed on any materials that are to contact the treatment site.

The study is intended to evaluate the large applicator of the Zeltiq Aesthetics non-invasive cooling device and to evaluate treatment of the lower abdomen to determine if non-invasive cold exposure will consistently result in a reduction of fat when used by clinicians in an environment that represents routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18 and 65 years of age.
* Clearly visible fat on an area of the lower abdomen appropriate for treatment with the non-invasive Zeltiq cooling device.
* Not had weight change fluctuations exceeding 5 pounds in the preceding 6 months.
* Read and sign a written informed consent form.

Exclusion Criteria:

* Had liposuction, or another surgical procedure(s) or mesotherapy (injections of minute natural extracts, drugs and other agents into the skin to eliminate fat deposits in cellulite) in area of intended treatment within the past 2 years.
* Had treatment with a cooling device within the past 6 months. (This exclusion does not apply to those enrolled in Group 3).
* Known history of injections into the abdomen (e.g., cortisone) within the past 6 months.
* Known history of cryoglobulinemia (abnormal blood proteins that thicken in cold temperatures), cold urticaria (large, allergic hives that occur when the skin is exposed to cold), or paroxysmal cold hemoglobinuria (sudden development of red blood cell breakdown causing hemoglobin [protein compound in blood] in the urine).
* Used diet pills within the past 6 months.
* Taking amino- or theophylline for asthma.
* You are unable or unwilling to comply with the study requirements.
* Any dermatological conditions or scars within the location of the treatment site that may interfere with the treatment or evaluation.
* Currently enrolled in a clinical study of any other unapproved investigational drug or device.
* Pregnant or intending to become pregnant in the next 9 months.
* Breastfeeding or have been breastfeeding in the past 9 months.
* Any other condition that would, in the professional opinion of the study doctor, potentially affect response or participation in this clinical study, or would pose an unacceptable risk to the subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 20 subjects, ages 18-65 years, who have clearly visible fat in the lower abdomen and are appropriate candidates as per the Study Doctor's physical examination.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-03; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy G Geronemus, MD, Principal Investigator — Laser & Skin Surgery Center of New York
Locations (1):
- Laser & Skin Surgery Center of New York, New York, New York, United States